CLINICAL TRIAL: NCT06182579
Title: Phase I Dose-Escalation Study of RiMO-401 With Radiation in Advanced Tumors
Brief Title: Phase I Study of RiMO-401 With Radiation in Advanced Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Coordination Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RiMO-401CL23-001
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor; Intratumoral Injection
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Intervention Model Description: dose escalation in a 3+3 study design
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RiMO-401 (Experimental): • Single intratumoral injection followed by radiation
  Interventions: Drug: RiMO-401

INTERVENTIONS:
Drug: RiMO-401 — • Single intratumoral injection of RiMO-401 followed by palliative radiotherapy
  Other Names: Radiation

SUMMARY:
This is a single arm study of RiMO-401 with radiation in patients with advanced tumors. A single escalation dose of RiMO-401 is intratumorally injected in a 3+3 study design to identify the recommended dose.

DETAILED DESCRIPTION:
Primary Objectives:

• To determine the tolerability of RiMO-401 with palliative radiation as assessed by CTCAEv5

Secondary Objectives:

* To determine clinical response of RiMO-401 with palliative radiotherapy
* To characterize adverse events of RiMO-401 in patients with advanced cancers
* To characterize the pharmacokinetics of RiMO-401 with palliative radiation

The target population comprises patients with clinically accessible lesions that can be trated with palliative radiation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced or metastatic cancer not amenable to curative therapy
* Lesion that is amenable to palliative radiotherapy
* Lesion that is technically feasible for intratumoral injection
* Target tumor in region not in the field that was irradiated within the past six months
* Patients with advanced or metastatic HNSCC must have progressed on or been intolerant to standard of care therapies including platinum-based chemotherapy and anti-PD(L)1 therapy, prior to study enrollment
* Patient must have recovered from acute toxic effects (≤ grade 1) of previous cancer treatments prior to enrollment
* Has measurable disease, defined as at least 1 tumor that fulfills the criteria for a target lesion
* ECOG score of 0-1
* Have a life expectancy of at least 12 weeks
* Have adequate bone marrow reserve and adequate liver function
* Both males and females and their partners of childbearing potential must agree to use adequate contraceptive measures
* Patients must sign a study-specific informed consent form prior to study entry
* Age 18 years or older.

Exclusion Criteria:

* Patients with a histological diagnosis of lymphomas and/or leukemias
* Patients with significant blood vessels (such as carotid artery encasement) or other major structures in the tumor region to be injected
* Patients may not have received chemotherapy, targeted therapies, immunotherapies, biologic response modifiers and/or hormonal therapy within the last 14 days
* Ongoing clinically significant infection at or near the incident lesion
* Major surgery over the target area (excluding placement of vascular access) <21 days from beginning of the study drug or minor surgical procedures <7 days
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that would make the patient inappropriate for enrollment in this study
* Has any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Pregnant and nursing women
* Patients with a target lesion located in a previously irradiated field
* Patients with a target lesion in the field that had complications from prior radiotherapy that are not amenable to repeat irradiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-06-16 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Determination of Recommended Dose | 45 Days
  The dose limiting toxicities of RiMO-401 with palliative radiation, as assessed by CTCAEv5, will not be observed in 33% or more patients

SECONDARY OUTCOMES:
Evaluation of Objective Response Rate (ORR) | 45 Days
  The Objective Response Rate (ORR) will be determined by imaging according to RECIST 1.1
Evaluation of Safety and Tolerability | 45 Days
  Incidence and severity of clinical and laboratory adverse events will be assessed according to CTCAEv5

OTHER OUTCOMES:
Evaluation of Maximum Plasma Concentration (Cmax) | 8 Days
  Plasma concentrations of RiMO-401 will be measured until 8 days after administration
Evaluation of Area Under the Curve (AUC) | 8 Days
  Plasma concentrations of RiMO-401 will be measured until 8 days after administration

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No